CLINICAL TRIAL: NCT04185506
Title: FReedom From Emotional Eating: Weight Loss Program
Brief Title: FReedom From Emotional Eating
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bowling Green State University (Other)
Responsible Party: Principal Investigator, Abby L. Braden, Ph.D., Assistant Professor, Bowling Green State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 879234-12
Record Dates: First submitted 2019-11-27; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Overweight and Obesity; Emotional Eating
Keywords: emotional eating; Dialectical Behavioral Therapy
MeSH Terms: conditions — Overweight; Obesity; Emotional Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DBT and behavioral weight loss (Experimental): The intervention is a 16-week group-based behavioral program consisting of a combination of Dialectical Behavioral Therapy (DBT) skills and behavioral weight loss techniques.
  Interventions: Behavioral: DBT+BWL

INTERVENTIONS:
Behavioral: DBT+BWL — DBT skills include a focus on emotion regulation, distress tolerance, and mindfulness techniques. BWL includes a focus on monitoring of food intake, calorie reduction, and dietary and physical activity education.

SUMMARY:
The current study was a pilot study examining a novel treatment for weight loss and emotional eating. The intervention is a group-based approach, and it includes a focus on teaching emotion regulation skills from Dialectical Behavioral Therapy and traditional behavioral weight loss techniques. The goal of the study was to develop and refine the treatment protocol. Additional goals of the study were to evaluate feasibility and acceptability, to see whether the intervention could be administered and whether participants like the treatment and believe it helps them. Changes in weight and emotional eating from baseline to post-treatment will also be measured.

DETAILED DESCRIPTION:
Background: The current study was a preliminary investigation of Live FREE, a pilot study of a treatment that included a combination of Dialectical Behavioral Therapy (DBT) and Behavioral Weight Loss (BWL) techniques for overweight/obese adult emotional eaters. Live FREE was based on the premise that impaired emotion regulation skills promote emotional eating behavior and lead to weight gain. Consistent with the ORBIT model (Czajkowski et al., 2015) of behavioral treatment development, the primary study aim was to refine the treatment protocol.

Methods: Adults with overweight/obesity who self-identified as emotional eaters were enrolled in Live FREE. Participants completed assessments at baseline, post-treatment, and at a 6-month follow-up. The intervention delivered 10-weeks of emotion regulation skills training followed by 6-weeks of BWL treatment in a group-based format. Groups were co-led by a licensed clinical psychologist and a doctoral student. Feasibility and acceptability will be examined by calculating rate of enrollment into the study and session attendance. ANOVA will be used to examine changes in primary and secondary outcome variables (weight, emotional eating) over time. Effect sizes (Cohen's d) will be calculated to examine the magnitude of change observed in these outcomes using standard interpretation guidelines ( d=0.2 be considered a 'small' effect size, 0.5 represents a 'medium' effect size and 0.8 a 'large' effect size).

ELIGIBILITY:
Inclusion Criteria:

* ability to read English at a 6th grade level
* willingness and ability to participate in study-related assessments and treatment visits. - - Subjects also had to report elevated levels of emotional eating. Elevated self-reported emotional eating occurred when subjects' self-reported emotional eating score was above the mean at least one of the sub scales of the Emotional Eating Scale (depression ≥ 21; EES-anxiety/anger ≥ 17; EES-boredom ≥ 21).

Exclusion Criteria:

* past or present medical condition that required physician monitoring to participate (i.e., history of coronary heart disease, hepatic disease, renal disease, stroke, seizures, or myocardial infarction; symptoms of angina; uncontrolled hypertension; diabetes; protein wasting disease/Cushing's syndrome; osteoarthritis; osteoporosis; orthopedic problems that would limit activity; or any other serious medical condition that would make physical activity unsafe)
* concurrent psychotherapy treatment
* concurrent enrollment in a weight loss program
* unstable dosage of psychotropic medication in the previous 3 months
* regular use of purging or other compensatory behaviors in the previous 3 months
* psychiatric conditions that would interfere with study participation (e.g., psychosis, current alcohol or drug use disorder, severe depression or suicidal behaviors within the past month)
* current use of weight altering medications (e.g., phentermine)
* immediate plans for weight loss surgery
* current pregnancy or breastfeeding.

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-04-16 (Actual); Primary Completion 2019-11-17 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
change in body weight | 10 months
  body weight measured in kilograms

SECONDARY OUTCOMES:
change in body mass index (BMI) | 10 months
  body weight in kilograms and height in meters will be used to calculate BMI (kg/m2)
change in emotional eating | 10 months
  Self-reported frequency of emotional eating is measured with the 25-item Emotional Eating Scale. Each item is scored on a 5-point scale ranging from 1 (no desire to eat) to 5 (overwhelming desire to eat). Total scores range from 25-125. Higher scores indicate more emotional eating.The Emotional Eating Scale yields 3 subscales: depression, anxiety/anger, and boredom.
change in emotion regulation | 10 months
  Self-reported difficulties in emotion regulation is measured with the 36-item Difficulties in Emotion Regulation Scale. Each item is scored on a scale ranging from 1 (almost never) to 5 (almost always). Ten items are reverse scored. Higher scores indicate more problems with emotion regulation. Total scores range from 36-180.
change in use of Dialectical Behavior Therapy (DBT) skills | 10 months
  The 38-item DBT skills subscale (DBT-WCCL-DSS) of the DBT Ways of Coping Checklist (DBT-WCCL) [37] is a self-report measure that assess DBT skills use. Items are scored on a scale ranging from 0 (never used) to 3 (regularly used). Higher scores indicate more frequent use of DBT skills. Total scores range from 0 - 114.